CLINICAL TRIAL: NCT05111288
Title: Influence of Pulse Electromagnetic Field Therapy on Myocardial Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney M. Wheatley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19-008996
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Exercise induced ischemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pulsed electromagnetic field (PEMF) therapy (Experimental): A portable PEMF device will be utilized. For the PEMF group, the device includes adjustable magnetic field strength range (X-axis: 0.22±0.05 mT, Y-axis: 0.20±0.05 mT and Z-axis: 0.06±0.02 mT) and working frequency (30±3Hz). This magnetic strength range and frequency will be maintained during 180 days of the study period. The subjects will be instructed to use their device three times per day: providing micromagnetic emitting on both hands (palms) during morning, afternoon and evening/night sessions. Each session takes 16 min (both hands, 8 min per hand) and thus subjects are exposed to therapy for 48 min per day. Subjects will use the device as outlined continuously up through the final days of testing.
  Interventions: Device: Pulsed electromagnetic field therapy (PEMF)
- Sham PEMF therapy (Sham Comparator): The sham PEMF devices are modified to deliver no micromagnetic field when turned on. The subjects will be instructed to use their device three times per day: providing micromagnetic emitting on both hands (palms) during morning, afternoon and evening/night sessions. Each session takes 16 min (both hands, 8 min per hand) and thus subjects are exposed to therapy for 48 min per day. Subjects will use the device as outlined continuously up through the final days of testing.
  Interventions: Device: Inactive Pulsed electromagnetic field therapy (PEMF)

INTERVENTIONS:
Device: Pulsed electromagnetic field therapy (PEMF) — Pulsed electromagnetic field (PEMF) therapy is a noninvasive technique, which provides low field electromagnetic stimulation. The therapy of PEMF is achieved by altering biological and physiological systems via low energy and non-ionizing electromagnetic fields.
  Arms: Pulsed electromagnetic field (PEMF) therapy
Device: Inactive Pulsed electromagnetic field therapy (PEMF) — PEMF device that turns on but does not provide any electromagnetic stimulation
  Arms: Sham PEMF therapy

SUMMARY:
This study is being done to observe the effects of treatment from a device called the Bioboosti which utilizes pulsed electromagnetic waves on its ability to improve blood flow to the heart tissue in individuals with coronary artery disease (CAD).

DETAILED DESCRIPTION:
Pulsed electromagnetic field (PEMF) therapy is a noninvasive technique, which provides low field electromagnetic stimulation. The therapy of PEMF is achieved by altering biological and physiological systems via low energy and non-ionizing electromagnetic fields. PEMF therapy was originally used clinically to manage osteoarthritis related pain and stiffness and to augment bone healing. In addition, recent research has explored the beneficial therapeutic effect of PEMF on microvasculature and circulation. More recently, research interest has been toward the effect of PEMF on various targets, including peripheral vascular function and blood flow. It has been suggested that PEMF therapy enhances the binding of free calcium (Ca2+) to calmodulin (CaM) and this phenomenon might improve tissue repair and pain and moreover other studies suggested an effect of PEMF on Ca/CaM-dependent nitric oxide (NO) signaling pathway, which is one of the major components for controlling vascular tone and blood pressure (BP, figure 1). The investigators have recently demonstrated that in subjects with metabolic syndrome with hypertension, 12 weeks of daily therapy using Bioboosti tended to lower BP and raise plasma NO levels as well as improve flow mediated dilation. In a small pilot study from China, subjects with a history of diffuse coronary disease and evidence of myocardial ischemia performed radionuclide SPECT before and after PEMF therapy or control. In this small pilot study there was evidence of reduced ischemia in the treatment group vs a control group. Thus the focus of this proposal is to pursue a larger clinical trial to demonstrate the benefits of PEMF therapy using the Bioboosti PEMF device to reduce the ischemic burden in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Known cardiac ischemia, who are non revascularizable, or have not and will not be undergo coronary intervention for the duration of their participation in the study.
* Evidence of ischemia from previous clinical tests (echo, nuclear, standard ECG from past 6 months).
* Left Ventricular Ejection fraction > 40% by echo (evaluated last 3 months).
* Able to complete a cardiopulmonary exercise test without significant non cardiac limitations, primarily orthopedic.
* On guideline directed optimal therapy for stable ischemia.

Exclusion Criteria:

* Anemia (< 7 mg/dl).
* Low potassium (< 3 mmol/L).
* Creatinine (> 5.0 mg/dl or < 0.6 mg/dl).
* Unable to exercise due primarily to orthopedic limitation.
* Severe lung disease.
* Morbid obesity (BMI > 42).
* Pregnant.
* Breast feeding.
* Significant arrhythmia (ventricular tachycardia, ventricular fibrillation, frequent premature ventricular contractions (PVCs), persistent atrial fibrillation, or 2nd or 3rd degree atrioventricular (AV) block).
* Seizures.
* Unstable angina.
* Coronary spasm.
* Recent myocardial infarction (< 90 days).
* Recent percutaneous coronary intervention (<90 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Myocardial blood flow during chemical stress | change from baseline to post 6 months treatment
  assessment of myocardial blood flow using 13N-ammonia myocardial perfusion positron emission tomography (PET) to quantify blood flow during chemical induced stress

SECONDARY OUTCOMES:
Peak Oxygen Consumption | change from baseline to post 6 months treatment
  Maximal oxygen consumption during maximal oxygen consumption
Seattle Angina Questionnaire | change from baseline to post 6 months treatment
  questionnaire to assess angina symptoms where scores range from 0- 100 and higher scores mean better outcomes or less angina symptoms
Time to angina onset during exercise | change from baseline to post 6 months treatment
  angina onset/threshold intensity during maximal exercise test
Exercise capacity (treadmill time) | change from baseline to post 6 months treatment
  total time on treadmill with maximal exercise test
New York Heart Association Heart Failure Functional classification | change from baseline to post 6 months treatment
  New York Heart Association classification on functional ability of heart failure patients based on symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Wheatley-Guy, PhD, Principal Investigator — Mayo Clinic; Bruce Johnson, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota